CLINICAL TRIAL: NCT03507972
Title: Evaluation of the Benefits of Ultrasound in Improving the Diagnosis and Management of the Child's Traumatic Ankle Injuries
Brief Title: Evaluation of the Benefits of Ultrasound in Improving the Diagnosis and Management of Injuries the Child's Ankle
Acronym: ANKLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: default inclusion
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014_35; 2015-A01127-42 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-01-15; First posted 2018-04-25 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Ankle Trauma
Keywords: ankle; diagnostic; ankle's ultrasound; traumatic lesion
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ankle ultrasound & ankle MRI (Other): Ankle ultrasound performed on the day of emergency consultation member MRI (without injection of contrast products) performed within 7 days following the trauma
  Interventions: Radiation: ankle ultrasound; Radiation: Member MRI

INTERVENTIONS:
Radiation: ankle ultrasound — Ankle ultrasound performed during emergencies visit.
Radiation: Member MRI — Member MRI (without injection of contrast product) performed within 7 days following the trauma

SUMMARY:
Evaluate ankle's ultrasound contribution in the accuracy of ankle's diagnosis of traumatic injuries (objectivated by reference's examination : ankle's MRI)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 5 years and < 18 years
* Isolated's trauma from one or both ankles
* First-line consultation for pediatrics emergencies at the University Hospital of Lille
* Informed and written consent of the holders of parental authority

Exclusion Criteria:

* Age < 5 years and ≥ 18 years
* History of trauma of the same ankle dating from less than 3 month
* History of surgery of this same ankle
* Constitutional or acquired bone disease
* Associated trauma affecting another anatomical region than the ankle or midfoot
* Polytrauma (presence of several traumas including at least one endangers vital functions)
* Associated wound requiring surgical exploration
* initial management of this trauma in another center
* Non affiliation to a social security scheme

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance rate of anatomical lesions of the ankle of ultrasound | Baseline (inclusion)
  Sensitivity of ankle ultrasound compared to MRI, considered as a gold standard, in the diagnosis of traumatic ankle injuries

SECONDARY OUTCOMES:
Diagnostic performance rate of anatomical lesions | Baseline (inclusion) and at visit 2 (within 7 days after the baseline)
  Specificity, predictive values (positive and negative) and likelihood ratios (positive and negative) of ultrasound versus MRI
The use of Ottawa decision rule | baseline (inclusion)
  the place of Ottawa criteria and ultrasound in the decision algorithm to limit standard radiographs (and thus irradiation).
  The Ottawa Ankle Rule was derived to aid in the efficient use of radiography in acute ankle and midfoot injuries.
orthopedic rehabilitation quality at 3 weeks according to the Oxford score. | at 3 weeks (control visit)
  The Oxford Ankle Foot Questionnaire for Children (OxAFQ-C) is used to measure subjective well-being for child patients (aged 5-16) affected by foot and ankle conditions using issues that are considered important to children.
  The OxAFQ-C has 15 items, 14 of which are used to calculate domain scores:
  Physical (6 items); School and Play (4 items) Emotional (4 items)

CONTACTS AND LOCATIONS:
Overall Officials: François Dubos, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Unité de pédiatrie Générale, Urgences et Maladies Infectieuses, Pôle de l'Urgence, Hôpital Roger Salengro, Lille, France

IPD SHARING:
Plan to Share IPD: No